CLINICAL TRIAL: NCT01389778
Title: Polycystic Ovary Syndrome Genetics and Treatment Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, Corrine Welt, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-P-002945
Record Dates: First submitted 2011-07-06; First posted 2011-07-08 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): Subjects treated with metformin.
  Interventions: Drug: Metformin ER; Drug: Metformin

INTERVENTIONS:
Drug: Metformin ER — Metformin ER 1500 mg for 12 weeks
Drug: Metformin

SUMMARY:
Polycystic ovary syndrome (PCOS) is the most common endocrine disorder in reproductive age women. Women with PCOS have a high risk of prediabetes, type 2 diabetes and heart disease. The investigators have found a possible change in the DNA (genes of the body that encode all of our traits) that seems to be related to insulin resistance. In this study, the investigators will try to determine whether the change in the gene affects a woman's ability to respond to a common treatment for PCOS, metformin.

These studies will uncover the change in a gene that might be one of the causes of PCOS. Discovering this gene will help better understand the diabetes and insulin abnormalities that are common in PCOS and will help us to better diagnose and treat PCOS to prevent the diabetes in these women.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS), which affects 7-10% of reproductive aged women, has traditionally been classified as a reproductive and dermatologic syndrome because of its high rate of infertility and the cosmetic complications of hyperandrogenism. However, it has become increasingly clear that insulin resistance is important in the pathogenesis of the disorder.

There are a number of variants that have been determined to be associated with PCOS risk. The investigators will determine the effect of these variants on the phenotype and response to treatment in PCOS. Subjects with PCOS will undergo extensive phenotyping including adipose tissue biopsy, dual energy X-ray absorptiometry (DXA, bone density) scan to examine adipose stores, an intravenous glucose tolerance test to study insulin sensitivity and beta cell function, androgen stimulation and inflammatory markers. The phenotyping will be repeated after 3 months of treatment with metformin. The studies will determine whether the genotype at PCOS risk variants dictates phenotype and response to treatment with metformin. Discovering genes involved in the etiology of PCOS will help pull us out of the endless circle that has characterized our understanding of PCOS pathophysiology for many years. The proposal also has the potential to illuminate one etiology of insulin resistance, which is present even in lean women with PCOS, and the impaired glucose tolerance and diabetes found in over 40% of PCOS patients.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome
* No medications for 1 month
* Good general health

Exclusion Criteria:

* Smoker
* Acute infection or chronic disease
* Diabetes
* Trying to get pregnant
* Bleeding disorders

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Insulin Sensitivity | 3 months

SECONDARY OUTCOMES:
Androgen Levels | 3 months
Ovulatory Rate | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Pau CT, Keefe C, Duran J, Welt CK. Metformin improves glucose effectiveness, not insulin sensitivity: predicting treatment response in women with polycystic ovary syndrome in an open-label, interventional study. J Clin Endocrinol Metab. 2014 May;99(5):1870-8. doi: 10.1210/jc.2013-4021. Epub 2014 Feb 25. PMID 24606093